CLINICAL TRIAL: NCT07037641
Title: Comparison of the Effectiveness of Chiropractic Manipulation Applied to the Lumbar Sacroiliac Region in Patients With Lumbar Disc Herniation
Acronym: CLuSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Asst. Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMT0008
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Spinal Manipulation; Chiropractic; Lumbal Disc Herniation
Keywords: Spinal Manipulation; Chiropractic; Lumbal Disc Herniation; Physiotherapy; Disc Pathology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this single-blind study, outcome assessments are conducted by an independent physiotherapist who is blinded to group allocation. The outcome assessor is not involved in the treatment sessions and does not have access to group assignment information. Participants and care providers are not blinded due to the nature of the manual interventions applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar Region Group (LBG) (Experimental): Participants in the lumbar manipulation group will receive the same conventional physiotherapy program as the control group (hot pack, TENS, ultrasound, and exercise therapy), along with high-velocity low-amplitude (HVLA) chiropractic manipulation applied specifically to the lumbar spine. The lumbar manipulation will be administered twice per week, totaling four sessions over a two-week period.
  Interventions: Other: Lumbar Spine Manipulation
- Sacroiliac Joint Manipulation Group (SEG) (Experimental): Participants in the sacroiliac joint manipulation group will receive the standard physiotherapy protocol (hot pack, TENS, ultrasound, and exercise therapy) in combination with high-velocity low-amplitude (HVLA) chiropractic manipulation targeted at the sacroiliac (SI) joint. The SI joint manipulation will be performed twice weekly, for a total of four sessions over two weeks.
  Interventions: Other: Sacroiliac Joint Manipulation
- Control Group (CG) (Active Comparator): Participants in the control group will receive conventional physiotherapy consisting of hot pack application, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound, and supervised exercise therapy. These treatments will be applied regularly over a two-week period. No chiropractic or manual therapy will be administered in this group.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Lumbar Spine Manipulation — Painful lumbar segments will be identified through palpation of the spinous and transverse processes. Patients will be positioned side-lying with head supported by a pillow. The lower arm will rest across the chest, and the lower leg will be extended while the upper leg will be flexed, with the foot placed in the popliteal space. The practitioner will assume a 45-degree angled stance, stabilizing the patient's pelvis between their thighs. The hypothenar eminence will contact the mammillary process of the dysfunctional vertebra, while the opposite hand stabilizes the upper shoulder. A high-velocity, low-amplitude (HVLA) thrust will be applied in a rotational direction toward the patient's umbilicus. This technique will be performed twice per week for two weeks (4 sessions total), alongside conventional physiotherapy (hot pack, TENS, ultrasound, and exercise).
  Arms: Lumbar Region Group (LBG)
Other: Sacroiliac Joint Manipulation — The side for sacroiliac joint manipulation will be determined using the Derifield leg length test. Based on functional leg length differences, a PI (posterior-inferior) ilium will be identified. Patients will be positioned side-lying with appropriate limb and trunk alignment. The practitioner's hypothenar eminence will be placed on the PSIS of the dysfunctional side. A high-velocity, low-amplitude (HVLA) thrust will be applied in a rotational direction from the PSIS toward the patient's umbilicus to correct the joint dysfunction. The manipulation will be performed twice a week over two weeks (4 sessions in total), combined with conventional physiotherapy (hot pack, TENS, ultrasound, and exercise).
  Arms: Sacroiliac Joint Manipulation Group (SEG)
Other: Conventional Physiotherapy — Conventional physiotherapy will consist of hot pack, TENS, therapeutic ultrasound, and supervised exercises applied over two weeks (6 sessions/week). Hot packs filled with silicate gel will be wrapped in four towel layers and applied for 20 minutes with the patient prone and a pillow under the abdomen. TENS will be delivered via Chattanooga Intelect device with a symmetrical biphasic program for 30 minutes using four electrodes placed on the treatment area. Ultrasound will be applied continuously for 3 minutes with the same device. Patients will be instructed on lumbar mobility and strengthening exercises, performed twice daily with 15 repetitions each. No spinal or sacroiliac manipulation will be performed in this group.
  Arms: Control Group (CG)

SUMMARY:
This study aims to compare the effectiveness of chiropractic manipulation applied to the lumbar and sacroiliac regions in patients with lumbar disc herniation. A total of 45 participants are randomly assigned into three groups (15 per group). The control group (CG) receives conventional physiotherapy, including hot pack, TENS, ultrasound, and exercise. The lumbar group (LG) receives the same physiotherapy program combined with lumbar spinal manipulation. The sacroiliac group (SIG) receives conventional physiotherapy combined with sacroiliac joint manipulation. Outcomes are measured using the Numeric Pain Rating Scale (NPRS), Quebec Back Pain Disability Scale, Tampa Scale for Kinesiophobia, and range of motion (ROM) assessments.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the comparative effectiveness of regional chiropractic manipulation in patients diagnosed with lumbar disc herniation. The study includes three groups, each consisting of 15 participants. All groups receive a standard physiotherapy protocol, including hot pack application, transcutaneous electrical nerve stimulation (TENS), therapeutic ultrasound, and exercise therapy.

The Control Group (CG) receives only the standard physiotherapy program. The Lumbar Group (LG) receives standard physiotherapy in combination with lumbar spinal manipulation.

The Sacroiliac Group (SIG) receives standard physiotherapy in combination with sacroiliac joint manipulation.

Interventions are delivered by licensed practitioners following standardized protocols. The study aims to evaluate the effects of region-specific chiropractic manipulations on pain intensity, functional disability, kinesiophobia, and lumbar range of motion. Assessments are conducted at baseline and at the end of the treatment period using validated measurement tools: the Numeric Pain Rating Scale (NPRS), Quebec Back Pain Disability Scale, Tampa Scale for Kinesiophobia, and goniometric range of motion measurements.

By comparing outcomes across these three groups, the study seeks to identify whether regionally targeted chiropractic manipulation enhances the clinical efficacy of conventional physiotherapy in managing lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65
* Have been diagnosed with lumbar disc herniation
* Have signed the voluntary consent form

Exclusion Criteria:

* Having a value below 4 according to the NAS
* Having a contraindication to chiropractic manipulation
* Having a rheumatic disease
* Having undergone surgery in the lumbar and sacroiliac regions
* Being pregnant or suspected of being pregnant
* Having a malignant disease
* Having severe physical and psychological disorders
* Having acute fractures of the spine and lower extremities fractures in the lower extremities
* Individuals with neurological and orthopedic deficits in the lower extremities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Numeric Pain Rating Scale - NPRS / NRS) | Baseline and at the end of 2 weeks
  Pain intensity will be assessed using the Numeric Pain Rating Scale (0-10), where higher scores indicate more severe pain.
Functional Disability (Quebec Back Pain Disability Scale) | Baseline and at the end of 2 weeks
  Functional disability due to low back pain will be measured using the Quebec Back Pain Disability Scale. Higher scores indicate greater disability.

SECONDARY OUTCOMES:
Kinesiophobia (Tampa Scale of Kinesiophobia - TSK) | Baseline and at the end of 2 weeks
  The Tampa Scale of Kinesiophobia will be used to assess fear of movement or re-injury. Higher scores indicate more severe kinesiophobia.
Lumbar Range of Motion (ROM) Measurements | Baseline and at the end of 2 weeks
  Lumbar flexion, extension, lateral flexion, and rotation will be measured using a goniometer to evaluate changes in spinal mobility.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA H HATIK, Asst. Prof., Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No